CLINICAL TRIAL: NCT02615067
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of 99mTc-MIP-1404 SPECT/CT Imaging to Detect Clinically Significant Prostate Cancer in Men With Biopsy Proven Low-Grade Prostate Cancer Who Are Candidates for Active Surveillance (proSPECT-AS)
Brief Title: Study to Evaluate 99mTc-MIP-1404 SPECT/CT Imaging in Men With Biopsy Proven Low-Grade Prostate Cancer
Acronym: proSPECT-AS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIP-1404-3301
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: Diagnostic; Active surveillance; Very low risk; Imaging; PSMA; SPECT/CT; 99mTc; Newly Diagnosed; Prostatectomy; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — technetium 99m 1-(1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)-2-((1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)methyl)-9,14-dioxo-2,8,13,15-tetraazaoctadecane-7,12,16,18-tetracarboxylic acid); lortalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 99mTc-MIP-1404 Injection (Experimental): 20 ± 3 millicurie (mCi) intravenous (IV) injection of 99mTc-MIP-1404
  Interventions: Drug: 99mTc-MIP-1404 Injection; Diagnostic Test: Whole-Body Planar and pelvic SPECT/CT scan

INTERVENTIONS:
Drug: 99mTc-MIP-1404 Injection — A single dose of 20 (±3) mCi intravenous (IV) injection of 99mTc-MIP-1404.
  Other Names: 1404
Diagnostic Test: Whole-Body Planar and pelvic SPECT/CT scan — A whole-body planar and pelvic SPECT/CT scan will be obtained 3-6 hours after injection of 99mTc-MIP-1404.

SUMMARY:
99mTc-MIP-1404 is a radioactive diagnostic imaging agent indicated for imaging men with newly diagnosed prostate cancer whose biopsy indicates a histopathologic Gleason Score of ≤ 3+4 severity who are candidates for active surveillance and are undergoing voluntary radical prostatectomy (RP) [Cohort A] or routine prostate biopsy [Cohort B]. This Phase 3 study is designed to evaluate the specificity and sensitivity of 99mTc-MIP-1404 SPECT/CT imaging to correctly identify subjects with previously unknown clinically significant prostate cancer.

DETAILED DESCRIPTION:
This is a multi-center, multi-reader, open-label trial, comparing 99mTc-MIP-1404 SPECT/CT imaging in men who have had a diagnostic trans-rectal ultrasound (TRUS) guided biopsy with a histopathologic finding of Gleason score ≤3+4 who are candidates for active surveillance and are undergoing routine biopsy or voluntary RP with or without a pelvic lymph node dissection (PLND). This study will evaluate the sensitivity and specificity of 99mTc-MIP-1404 SPECT/CT image assessments to correctly identify subjects with previously unknown clinically significant prostate cancer in two cohorts: (1) Low grade prostate cancer who have elected to undergo RP [Cohort A]; and (2) very low risk (VLR) prostate cancer per 2016 NCCN Guidelines who are scheduled to undergo routine prostate biopsy [Cohort B].

Subjects will receive a single dose of 99mTc-MIP-1404 Injection (study drug) followed by whole body planar and SPECT/CT (pelvic) imaging 3-6 hours after injection. In accordance with standard of care procedures, subjects will undergo either voluntary RP [Cohort A] or prostate biopsy [Cohort B] within 42 days after study drug dosing. 99mTc-MIP-1404 image data will be collected by a central imaging core laboratory and evaluated for visible uptake within the prostate gland. These findings will then be compared against central histopathology as the truth standard. The central imaging core lab independent readers for the SPECT/CT scans will be blinded to all clinical data, including pathology results. Likewise, central pathologists are to remain blinded to all clinical data, including imaging results.

ELIGIBILITY:
INCLUSION CRITERIA:

* Ability to provide informed consent and willingness to comply with protocol requirements
* Life expectancy ≥ 6 months

Cohort A only:

* A diagnostic trans-rectal ultrasound (TRUS)-guided biopsy within 12 months of enrollment showing adenocarcinoma of the prostate gland
* Within 90 days of consent, serum PSA ≤ 15.0 ng/mL or ≤ 7.5 ng/mL if on 5 α-reductase inhibitors.
* Candidates for active surveillance and/or a Gleason score ≤3+4
* Scheduled to undergo radical prostatectomy (RP) with or without pelvic lymph node dissection (PLND)

Cohort B only:

* Very low risk (VLR) prostate cancer defined by 2016 NCCN Guideline criteria:
* T1c stage, and
* PSA < 10 ng/mL, and
* Gleason score ≤ 6 with < 3 biopsy cores cancer positive and ≤ 50% cancer in any core based on prior prostate biopsy within 24 months of enrollment, and
* PSA density < 0.15 mg/mL/g
* Scheduled to undergo a reassessment of prostate cancer staging that includes prostate biopsy as part of routine follow-up

EXCLUSION CRITERIA:

1. Subjects administered a radioisotope within 5 physical half-lives prior to study drug injection.
2. Previous treatment with hormonal therapy, surgery (except biopsy), radiation therapy, LHRH analogs, and non-steroidal anti-androgens, for the treatment of prostate cancer or benign prostatic hyperplasia (BPH)
3. Planned androgen or anti-androgen therapy prior to RP surgery or biopsy
4. Subjects with any medical condition or other circumstances that, in the opinion of the investigator, would significantly interfere with obtaining reliable data, achieving study objectives, or completing the study
5. Malignancy (not including curatively treated basal or squamous cell carcinoma of the skin) within the previous 5 years. (Ta stage transitional cell carcinoma bladder cancer with negative surveillance cystoscopy within the past 2 years may be included).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Specificity of 99mTc-MIP-1404 to detect clinically significant prostate cancer when compared to histopathology following either RP [Cohort A] or prostate biopsy [Cohort B] | Within 3-6 hours of dosing, SPECT/CT and whole body planar images will be taken
  Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of the prostate and pelvic lymph nodes, if applicable, (as determined by histopathology) in patients undergoing RP (with or without extended pelvic lymph node dissection) or routine prostate biopsy. Pathology results will be used as the truth standard for all imaging analyses.
Sensitivity of 99mTc-MIP-1404 to detect clinically significant prostate cancer when compared to histopathology following either RP [Cohort A] or prostate biopsy [Cohort B] | Within 3-6 hours of dosing, SPECT/CT and whole body planar images will be taken
  Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of the prostate and pelvic lymph nodes (as determined by histopathology) in patients undergoing standard of care prostatectomy with or without extended pelvic lymph node dissection. Pathology results will be used as the truth standard for all imaging analyses.

SECONDARY OUTCOMES:
Sensitivity of 99mTc-MIP-1404 in prostate segments as compared to histopathology following RP [Cohort A only] | Within 3-6 hours of dosing, SPECT/CT and whole body planar images will be taken
  Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of the prostate (as determined by histopathology)
Specificity of 99mTc-MIP-1404 in prostate segments as compared to histopathology following RP [Cohort A only] | Within 3-6 hours of dosing, SPECT/CT and whole body planar images will be taken
  Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of the prostate (as determined by histopathology)
Clinical safety of 99mTc-MIP-1404 | Changes in vital signs and clinical laboratory test results from time of screening until pre-surgery (Day 0 - 42). Treatment-emergent adverse events from study drug injection until pre-surgery or pre-biopsy (within 42 days)
  Clinical laboratory tests will include hematology and clinical chemistry. Vital signs will include heart rate, blood pressure, temperature and respiration rate.

CONTACTS AND LOCATIONS:
Overall Officials: William Ellis, MD, Study Chair — University of Washington
Locations (45):
- United States (33):
  - City of Hope Cancer Center, Duarte, California
  - VA Greater Los Angeles Healthcare, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Urology Partners - Tampa Bay, Clearwater, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - University of Georgia / Regents Medical Center, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Montgomery General Hospital, Olney, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cooper Health System, Camden, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Northeast Urology Research, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Urologic Consultants of Southeastern PA, LLP, Bala-Cynwyd, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Rockledge, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (12):
  - Prostate Cancer Centre, Calgary, AB, Alberta
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Cancer Care Nova Scotia, Halifax, Nova Scotia
  - Ottawa Hospital Research Institute, University of Ottawa, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - MUHC, Montreal, Quebec
  - Centre d'imagerie moléculaire de Sherbrooke, Sherbrooke, Quebec
  - Hôtel-Dieu de Québec, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vallabhajosula S, Nikolopoulou A, Babich JW, Osborne JR, Tagawa ST, Lipai I, Solnes L, Maresca KP, Armor T, Joyal JL, Crummet R, Stubbs JB, Goldsmith SJ. 99mTc-labeled small-molecule inhibitors of prostate-specific membrane antigen: pharmacokinetics and biodistribution studies in healthy subjects and patients with metastatic prostate cancer. J Nucl Med. 2014 Nov;55(11):1791-8. doi: 10.2967/jnumed.114.140426. Epub 2014 Oct 23. PMID 25342385
- [Background] Eder M, Eisenhut M, Babich J, Haberkorn U. PSMA as a target for radiolabelled small molecules. Eur J Nucl Med Mol Imaging. 2013 Jun;40(6):819-23. doi: 10.1007/s00259-013-2374-2. No abstract available. PMID 23463331
- [Background] Hillier SM, Maresca KP, Lu G, Merkin RD, Marquis JC, Zimmerman CN, Eckelman WC, Joyal JL, Babich JW. 99mTc-labeled small-molecule inhibitors of prostate-specific membrane antigen for molecular imaging of prostate cancer. J Nucl Med. 2013 Aug;54(8):1369-76. doi: 10.2967/jnumed.112.116624. Epub 2013 Jun 3. PMID 23733925